CLINICAL TRIAL: NCT02662894
Title: Efficacy of Fixed-dose Combination of Valsartan + Rosuvastatin Versus Their Isolated Components for Hypertension and Dyslipidemia.
Brief Title: Fixed-dose Combination of Valsartan + Rosuvastatin Versus Their Isolated Components for Hypertension and Dyslipidemia.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMS0815
Record Dates: First submitted 2015-11-23; First posted 2016-01-26 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Valsartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Valsartan 160mg + Rosuvastatin 20mg (Experimental): Fixed-dose combination of valsartan (160mg) + rosuvastatin (20 mg), oral, once daily.
  Interventions: Drug: Valsartan 160mg + Rosuvastatin 20mg
- Valsartan 320mg + Rosuvastatin 20mg (Experimental): Fixed-dose combination of valsartan (320 mg) + rosuvastatin (20 mg), oral, once daily.
  Interventions: Drug: Valsartan 320mg + Rosuvastatin 20mg
- Diovan® 160mg + Crestor® 20mg (Active Comparator): Take together 1 tablet of Diovan (160mg) plus 1 tablet of Crestor (20mg), oral, once daily.
  Interventions: Drug: Diovan® 160mg + Crestor® 20mg
- Diovan® 320mg + Crestor® 20mg (Active Comparator): Take together 1 tablet of Diovan (320mg) plus 1 tablet of Crestor (20mg), oral, once daily.
  Interventions: Drug: Diovan® 320mg + Crestor® 20mg

INTERVENTIONS:
Drug: Valsartan 160mg + Rosuvastatin 20mg — 1 tablet, oral, a day
  Arms: Valsartan 160mg + Rosuvastatin 20mg
Drug: Valsartan 320mg + Rosuvastatin 20mg — 1 tablet, oral, a day
  Arms: Valsartan 320mg + Rosuvastatin 20mg
Drug: Diovan® 160mg + Crestor® 20mg — Take together 1 tablet of Diovan (160mg) plus 1 tablet of Crestor (20mg), oral, once daily.
  Other Names: Valsartan 160mg + Rosuvastatin 20mg
  Arms: Diovan® 160mg + Crestor® 20mg
Drug: Diovan® 320mg + Crestor® 20mg — Take together 1 tablet of Diovan (320mg) plus 1 tablet of Crestor (20mg), oral, once daily.
  Other Names: Valsartan 320mg + Rosuvastatin 20mg
  Arms: Diovan® 320mg + Crestor® 20mg

SUMMARY:
Noninferiority trial to assess efficacy of fixed-dose combination of valsartan + rosuvastatin versus their isolated components in treatment of hypertension and dyslipidemia.

DETAILED DESCRIPTION:
* Open-label,randomized, multicenter;
* Maximal experiment duration: 8 weeks;
* 04 visits;
* Safety and efficacy evaluation

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes aged between 18 and 65 years;
* Participants diagnosed with uncontrolled hypertension;
* Participants with intermediate and high risk dyslipidemia, according to the V Brazilian Guidelines on Dyslipidemia and Prevention of Atherosclerosis;
* Ability to understand and consent to participate in this clinical study, manifested by signing the Informed Consent and Informed ( IC) .

Exclusion Criteria:

* Participants with a previous diagnosis of familial hypercholesterolemia (homozygous);
* Concomitant use of angiotensin II receptor blocker (ARB) or inhibitor of angiotensin converting enzyme (ACE);
* participants with isolated hypertriglyceridemia (TG ≥150 mg / dL) according to V Brazilian Guidelines on Dyslipidemia and Prevention of Atherosclerosis;
* research participants with total cholesterol (TC) above 500 mg / dL or triglyceride (TG) above 400 mg / dL;
* participants with systolic blood pressure ≥180 mmHg or diastolic ≥110 mmHg;
* research participants with postural hypotension (SBP decrease ≥20 mmHg or DBP ≥10 mmHg in orthostatic position in relation to the sitting position);
* History of congestive heart failure (CHF) functional class III or IV (NYHA);;
* any clinical, laboratory and electrocardiographic that, in the judgment of the investigator, may interfere with the safety of research participants;
* Creatine phosphokinase (CPK) levels above the established laboratory normal range;
* Transaminases (ALT and ASL) serum above 2 times the established laboratory normal range;
* Body mass index (BMI) ≥35 kg / m²;
* Immunocompromised participants (eg .: malignancies, patients with Acquired Immunodeficiency Syndrome etc);
* Chronic use of drugs that may interact with the drugs of the study;
* Patients on concomitant lipid-lowering therapy;
* History hypersensitivity to the active ingredients used in the study;
* Participants who are pregnant, nursing or planning to become pregnant, or female participants of childbearing potential who are not using a reliable method of contraception;
* History of alcohol abuse or illicit drug use;
* Adherence to uniformization medication <80%;
* Participating in the research that has participated in clinical trial protocols in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, sub-item J), unless the investigator considers that there may be direct benefit to it;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of systemic blood pressure measured between the first visit and last visit. | 8 weeks
Percentage of participants who reach the goal of LDL-C according to intermediate risk rating ( LDLc < 100mg / dL ) and high risk ( LDLc < 70 mg / dL ) . | 8 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded after the signing of the Informed Consent ( IC) and until the end of the study. | 8 weeks